CLINICAL TRIAL: NCT01452282
Title: Ankle-Brachial Index Estimating Cardiac Complications After Non-Cardiac Surgery
Brief Title: Ankle-Brachial Index Estimating Cardiac Complications After Surgery
Acronym: ABRACOS
Status: Completed | Type: Observational
Sponsor: University of Sao Paulo (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Principal Investigator, Bruno Caramelli, Director, Interdisciplinary Medicine in Cardiology Unit, Heart Institute, University of Sao Paulo
Other Study IDs: USP - 0175/11
Record Dates: First submitted 2011-10-08; First posted 2011-10-14 (Estimated); Last update posted 2013-11-13 (Estimated); Status verified 2013-11

CONDITIONS: Cardiovascular Complications; Myocardial Infarction; Acute Coronary Syndromes
Keywords: Ankle Brachial Index; Perioperative care; General Surgery; Acute Coronary Syndromes; Cardiovascular Complications
MeSH Terms: conditions — Myocardial Infarction; Acute Coronary Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Whole blood samples will be retained for future exams.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Ankle Brachial Index

SUMMARY:
Introduction: Patients undergoing noncardiac surgery are at increased risk of cardiovascular complications. The development of methods that can accurately predict the occurrence of these events is of critical importance and large studies have been published with this purpose. Based on these studies, several algorithms have been proposed to predict of cardiovascular events postoperatively. However, quantification of this risk is often difficult to measure, especially in those patients with subclinical disease, not always detected in routine evaluation. The ankle brachial index (ABI) has proved a valuable tool in the quantification of cardiovascular risk, and perhaps the most promising when compared with other methods. It is easy, cheap, fast and feasible in office care, with a great acceptance between patients and small intra and inter observer variability. Despite strong evidence of the utility of ABI as a tool in assessing cardiovascular risk, there are no data about the use of ABI in other patients referred for non vascular surgery, which constitutes the majority of operations performed worldwide.

Objectives: To evaluate the use of ABI as a predictor of cardiovascular events in patients undergoing non-cardiac and non-vascular surgery and its applicability as a tool in the reclassification of patient risk groups established by guidelines for perioperative evaluation.

Methods: 300 moderate to high risk patients referred for non-vascular and non-cardiac will be included. Data about risk factors, signs and symptoms, physical examination and treatment used will be collected before surgery. The ABI will be measured and the patient will be monitored for 30 days to the detection of cardiovascular events: death from any cardiovascular causes, unstable angina, nonfatal myocardial infarction, isolated elevation of troponin, decompensated heart failure, cardiogenic shock, stop nonfatal heart failure, pulmonary edema, stroke and lower limb ischemia. Postoperative electrocardiogram, total creatine kinase, MB fraction and troponin I will be measured daily until 3º day and whenever clinically indicated.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 or older, moderate to high risk by Revised Cardiac Risk and the Modified Cardiac Risk Index undergoing non-cardiac and non-vascular surgery will be referred for the study.

Exclusion Criteria:

* Patients with atrial fibrillation, aortic regurgitation, low risk of cardiovascular complications by the Revised Cardiac Risk and the Modified Cardiac Risk Index and those referred for vascular or cardiac surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Both sex patients aged 18 or older, undergoing non-cardiac and non-vascular surgery will be referred for the study.
Sampling Method: Non-Probability Sample
Enrollment: 196 (Actual)
Dates: Start 2011-10; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Major Cardiovascular Events | 30 days after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Bruno Caramelli, Ph.D., Principal Investigator — Heart Institute - University of Sao Paulo; Gabriel A Carmo, M.D., Principal Investigator — Heart Institute - University of Sao Paulo
Locations (1):
- University of Sao Paulo, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Carmo GA, Calderaro D, Gualandro DM, Pastana AF, Yu PC, Marques AC, Caramelli B. The Ankle-Brachial Index is Associated With Cardiovascular Complications After Noncardiac Surgery. Angiology. 2016 Feb;67(2):187-92. doi: 10.1177/0003319715589684. Epub 2015 Jun 9. PMID 26058673